CLINICAL TRIAL: NCT01158586
Title: Postoperative Patient Controlled Epidural Analgesia After Total Knee Arthroplasty With 2ug/ml Fentanyl Combine With 0.2% Ropivacaine or 0.2% Levobupivcaine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: United Christian Hospital (Other)
Responsible Party: Dr. Anthony Kui Hung Njo, Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCEA-LEVO-ROPI
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-02

CONDITIONS: Arthroplasty, Replacement, Knee; Patient-controlled Analgesia
Keywords: post total knee replacement; patient control; epidural analgesia
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levobupivacaine (Experimental): patient control epidural analgeisa using 0.2% levobupivacaine with 2ug/ml fentanyl
  Interventions: Drug: Levobupivacaine
- Ropivacaine (Active Comparator): patient controlled epidural analgesia using 0.2% ropivacaine with 2ug/ml fentanyl
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — patient control epidural analgesia using 0.2% levobupivacaine with 2ug/ml fentanyl

SUMMARY:
Postoperative epidural analgesia (EA) is an effective and well-accepted modality of pain relief technique after having total knee replacement operation(1,4). Patient controlled epidural analgesia (PCEA) has been shown to be safe and effective in standard ward setting(2) and results in reduced epidural analgesic requirements(3). Besides, it also bear the advantage of avoidance of overdose, reduction of waiting times and involvement of patients in their analgesic regimen(3). Both ropivacaine and levobupivacaine are the local anaesthetic using in epidural analgesia which has been proven to be safe and effective(4). 0.2% Ropivacaine with 2ug/ml fentanyl has been used in our locality for more than 8 years. Another local anaesthetics, levobupivacaine, a S-enantiomer of bupivacaine has come up in Hong Kong, which has been proved to be safe, effective and may be better value for money. These two drugs has been proven to have similar analgesic potency in using as EA for postoperative pain relief for other operation(5,6,7) and for orthropaedics operation but in different concentration(4). Concerns have been raised about the introduction of the levobupivacaine in the departmental protocol. Objectives of this study are A)to determine the equivalence of two local anaesthetics regimen ; 0.2% ropivacaine with 2ug/ml fentanyl and 0.2% levobupivacaine with 2ug/ml fentanyl and B) to assess the cost-effectiveness of using these two regimens.

The null hypothesis is that the difference of analgesic effect, presented with visual analogue score, of two patient controlled epidural analgesia regimen, the 0.2% ropivacaine with 2 ug/ml fentanyl and 0.2% levobupivacaine with 2ug/ml fentanyl is higher than the threshold of 9 mm VAS. (8,9,10)

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old, ASA I -III and
* Undergoing total knee arthroplasty
* Combine spinal-epidural anaesthesia

Exclusion Criteria:

* Known hypersensitivity to amide-type local anaesthetics
* Known hypersensitivity to opioids
* Known history of severe cardiovascular, renal, hepatic, neurological or psychiatric disease as judged by the investigator
* Known history of peripheral neuropathies
* Those receiving chronic analgesic therapy, or any contraindication for epidural analgesia (e.g. clotting disorders, or history of lumbar surgery)
* Inability to perform a pain score, or pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Pain score | 48hours after start epidural analgesia
  as well as complications from epidural analgesia are also going to record and monitored

SECONDARY OUTCOMES:
cost/treatment | 48hours

CONTACTS AND LOCATIONS:
Locations (1):
- United Christian Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Reference 1. Block et al. Efficiancy of postoperative epidural analgesia: A meta-analysis. JAMA 290: 2455-63 2. Werawatganon T. Patient controlled intravenous opioid analgesia versus continuous epidural analgesia for pain after intra-abdominal surgery. The Cochrane Databas of systemic reviews. Issue 3 Art. No.: No.: CD 004044. DOI: 10.1002/14651858. CD004088.pub2. 3. Liu SS et al. Patient-controlled epidural analgesia with bupivacaine and fentanyl on hospital wards: propective experience with 1,030 surgical patients Anesthesiology 88: 388-95 4. Silvasti M et al. Patient-controlled analgesia versus continuous epidural analgesia after total knee arthroplasty Acta Anaesthesiol Scand 42: 576 - 80 5. Stand T et al. Patient-controlled epidural analgesia reduces analgesic requirements compared to continuous epidural infusion after major abdominal surgery. Can J Anaesth 50:258-64 6. Linda S. et al. Relative Analgesic Potencies of Levobupivacaine and Ropivacaine for Epidural Analgesia in Labor. Anesthesiology 2003; 99:1354-8 7. Marc Senard et al. Epidural Levobupivacaine 0.1% or Ropivacaine 0.1% Combined with Morphine Provides Comparable Analgesia After Abdominal Surgery Anesth Analg 2004;98:389-94 8. Kelly AM The minimum clinically significant difference in visual analogue scale pain score does not differ with severity of pain.Emerg Med J 2001; 18:205-07 9. Mark MSM et al. The minimum clinically significant difference in visual analogue scale pain score in a local emergency setting. Hong Kong Journal of Emergency Medicine 2009; 16(4): 234-6 10. Kelly AM. Does the clinically significant difference in visual analog scale pain scores vary with gender, age, or cause of pain? Acad Emerg Med. 1998 Nov; 5(11): 1086-90.